CLINICAL TRIAL: NCT01611298
Title: Transfer of Donor-Derived Humoral Immunity Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Donor-Derived Humoral Immunity, Hematopoietic Stem Cell Transplantation, TAR
Acronym: TAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Krance (Other)
Collaborators: Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Robert Krance, Prof, Pediatrics-Hema & Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-21942-TAR
Record Dates: First submitted 2012-04-11; First posted 2012-06-04 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Hodgkin Lymphoma; Non-Hodgkin Lymphoma
Keywords: allogeneic stem cell transplant; malignant diseases; Acute lymphoblastic leukemia; acute myelogenous leukemia; Chronic myelogenous leukemia; myelodysplastic syndrome; Hodgkin lymphoma; non-Hodgkin lymphoma; myeloproliferative disorder; non-malignant disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myeloproliferative Disorders | interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm: Tetanus Toxoid (Experimental): SCT Donors will receive one dose of tetanus toxoid 0.5mL intramuscularly into deltoid or medial lateral thigh 7-10 days prior to bone marrow or peripheral blood stem cell harvest
  Interventions: Biological: Tetanus

INTERVENTIONS:
Biological: Tetanus — Stem cell transplant donors will receive one dose of tetanus toxoid 0.5mL intramuscularly into deltoid or medial lateral thigh 7-10 days prior to bone marrow or peripheral blood stem cell harvest.
  Stem cell transplant recipients will receive one dose of tetanus toxoid 0.5mL intramuscularly (or subcutaneously if platelet count less than 50,000/uL) into deltoid or medial lateral thigh 7-10 days prior to stem cell transplant (FIRST dose).
  Stem cell transplant recipients will receive a subsequent dose of tetanus toxoid 0.5mL given intramuscularly into deltoid or medial lateral thigh (or given subcutaneously if platelet count is less than 50,000/uL) approximately 3 months following allo stem cell transplant. Patients must meet re-evaluation criteria to receive injection.
  Other Names: Tetanus Toxoid vaccine

SUMMARY:
This research study is for subjects that are receiving a bone marrow transplant. As part of the transplant subjects will receive stem cells from a donor who has agreed to donate stem cells for them. Unfortunately, it takes a long time for the immune system to recover after a bone marrow transplant. This makes it more likely for patients to develop serious infections.

This study is being done to better understand how the immune system will recover after transplant. The immune system includes the cells that help fight infection. This study will help investigators understand which patients are at risk for developing infections after transplant.

All children and adults receive standard vaccines (shots) during their lifetime to provide protection from many different infections. One such infection is tetanus, a bacteria that can cause life-threatening problems. After transplant patients no longer have protection from infections such as tetanus. Therefore, most patients need to receive all their vaccine (shots) again after transplant. This is usually done 1-2 years after transplant, since it may take that long for patients to have a normal immune system.

However, the investigators believe that the time it will take for the patient to develop normal protection against tetanus can be shortened if both the patient and the patient's stem cell donor receive a tetanus vaccine.

The goal of this study is to determine if giving a tetanus vaccine to the donor and the patient will provide the patient with enough protection (immunity) to prevent infection following bone marrow transplant.

DETAILED DESCRIPTION:
To participate in this study, patients will need to have given informed consent to have a bone marrow transplant. Before receiving the tetanus vaccine, we would like to test the patient's immune system against tetanus. We will again want to test the patient's immune system against tetanus on the day the patient receives the bone marrow transplant. Approximately 3 months after transplant, if the patient is still eligible, they will receive an additional tetanus booster shot. We will again draw blood to test their immune system against tetanus at the time points listed below.

TREATMENT PLAN:

If the subject meets eligibility requirements and consents to be part of this study, we will collect 8 mL (1.7 teaspoons) of blood from the subject to test their immunity 7 to 10 days before their bone marrow transplant. The subject will receive a tetanus vaccine (given as an injection into the upper arm or thigh muscle) on that same day. We will then collect approximately the same amount of blood (2 teaspoons) on the day the patient would receive the bone marrow transplant. We will also collect the same amount of blood 1 week, 2 weeks, 4 weeks and 3 months, 6 months and 12 months after the transplant. This will help us to see how the patients immune system responded to the vaccine.

Three months after the transplant, the patient will receive an additional tetanus vaccine (known as a booster shot), but only if the patient is still eligible to receive it. Patient's will only be eligible to receive the booster shot if they remain well and do not have any other problems such as severe infection, graft versus host disease or relapse. We will collect 8 ml (1.7 teaspoons) of blood 1 week, 2 weeks and 4 weeks after receiving the booster shot to determine if they respond to the vaccine.

ELIGIBILITY:
INCLUSION CRITERIA:

Inclusion Criteria for Donors:

* Related donor of bone marrow or peripheral blood stem cell product
* Age 3 to 70 years
* Informed consent form signed and sent to Research Coordinator

Inclusion Criteria for Recipients:

* Patient with acute lymphoblastic leukemia, acute myelogenous leukemia, chronic myelogenous leukemia, myelodysplastic syndrome, myeloproliferative disorder, Hodgkin lymphoma, non-Hodgkin lymphoma, or a non-malignant disease requiring allogeneic stem cell transplant
* Age between 3 and 70 years
* Informed consent form signed and sent to Research Coordinator

EXCLUSION CRITERIA:

Exclusion Criteria for Donors:

* Allergy to tetanus vaccine
* Pregnant or lactating
* Has received tetanus booster within preceding 12 months

Exclusion Criteria for Recipients to Receive FIRST Tetanus Immunization:

* Allergy to tetanus vaccine
* Has received tetanus booster within preceding 12 months
* Has active malignancy (not in remission)

Exclusion Criteria for Recipients to Receive SUBSEQUENT Tetanus Immunization:

* Allergy to tetanus vaccine
* Active, acute graft vs. host disease (GVHD) greater than or equal to grade II or chronic graft vs. host disease (GVHD)
* Disease relapse - less than 75% donor chimerism (peripheral blood or bone marrow)
* Active infection (bacterial, viral, fungal) or fever (temperature greater than 100.5 celsius)

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-03; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krance, MD, Study Director — Texas Childrens Hospital / Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Childen's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Tetanus Toxoid: SCT Donors will receive one dose of tetanus toxoid 0.5mL intramuscularly into deltoid or medial lateral thigh 7-10 days prior to bone marrow or peripheral blood stem cell harvest
  Tetanus: Stem cell transplant donors will receive one dose of tetanus toxoid 0.5mL intramuscularly into deltoid or medial lateral thigh 7-10 days prior to bone marrow or peripheral blood stem cell harvest.
  Stem cell transplant recipients will receive one dose of tetanus toxoid 0.5mL intramuscularly (or subcutaneously if platelet count less than 50,000/uL) into deltoid or medial lateral thigh 7-10 days prior to stem cell transplant (FIRST dose).
  Stem cell transplant recipients will receive a subsequent dose of tetanus toxoid 0.5mL given intramuscularly into deltoid or medial lateral thigh (or given subcutaneously if platelet count is less than 50,000/uL) approximately 3 months following allo stem cell transplant. Patients must meet re-evaluation criteria to receive injection.
Period: Overall Study
Arm/Group | Single Arm: Tetanus Toxoid
Started | 7
Completed | 5
Not Completed | 2
Not completed — Relapsed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Tetanus Toxoid
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 7 [3 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1
  White | 6
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Antibody Recall Response Rate
Description: The proportion of participants with antibody recall response along with 95% confidence intervals will be calculated.
Time Frame: 4 months
Population: One participant was off study on day 68 and not included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Single Arm: Tetanus Toxoid
Number analyzed (Participants) | 6
proportion of participants | 0.167 [0.004 to 0.641]

2. Secondary Outcome: Change in Immunoglobulin Levels
Description: Changes from baseline to several time points during follow-up will be calculated.
Time Frame: up to 12 months
Population: One participant was off study on day 68 and not included in this analysis. Six participants included in the analysis had at least one measurement at the follow-up time points. n=the number of participants with measurements for that time point.
Measure: Median (Inter-Quartile Range); unit: MG/DL
Arm/Group | Single Arm: Tetanus Toxoid
Number analyzed (Participants) | 6
MG/DL
  IgA Change at 3 months: number analyzed (Participants) | 5
  IgA Change at 3 months | -49.9 [-68.0 to -31.0]
  IgA Change at 6 months: number analyzed (Participants) | 3
  IgA Change at 6 months | -1.0 [-29.0 to 66.0]
  IgA Change at 12 months: number analyzed (Participants) | 5
  IgA Change at 12 months | 7.7 [-34.0 to 16.0]
  IgG Change at 3 months: number analyzed (Participants) | 5
  IgG Change at 3 months | -677.6 [-717.0 to -676.1]
  IgG Change at 6 months: number analyzed (Participants) | 3
  IgG Change at 6 months | -668.2 [-678.0 to -369.0]
  IgG Change at 12 months: number analyzed (Participants) | 5
  IgG Change at 12 months | -683.0 [-1182.0 to -659.5]
  IgM Change at 3 months: number analyzed (Participants) | 5
  IgM Change at 3 months | 13.7 [11.9 to 30.5]
  IgM Change at 6 months: number analyzed (Participants) | 3
  IgM Change at 6 months | 45.0 [21.6 to 148.0]
  IgM Change at 12 months: number analyzed (Participants) | 5
  IgM Change at 12 months | 75.8 [40.0 to 98.0]

ADVERSE EVENTS:
Time Frame: Toxicities will be assessed while patients are receiving tetanus toxoid and for 6 weeks following last vaccination, either 6 weeks after the first booster or 6 weeks after the second booster, if the patient receives the second booster.
Description: All adverse events were collected using CTCAE 3.0 for the study. For reporting purpose, adverse event terms were converted using CTCAE v4.0.
Arm/Group | Single Arm: Tetanus Toxoid
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Tetanus Toxoid (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infection - Other: Gastrointestinal Abdomen (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Tetanus Toxoid (N=7)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (11)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 6 (22)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (21)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 4 (11)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (2)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (22)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Mucosal infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Febrile neutropenia(fever of unknown origin wo clinically or microbiologically documented infection) (Blood and lymphatic system disorders) | 2 (2) — ANC < 1.0x10e9/L,fever >=38.5 degrees C
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (5)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 3 (8)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (7)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (3)
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection(documented clinically or microbiologically) with Grade 3 or 4 neutrophils-Bladder(urinary) (Infections and infestations) | 1 (1) — ANC <1.0 x 10e9/L
Infection - Other: Mucosa (Infections and infestations) | 1 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1)
Lipase (Investigations) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (21)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 4 (10)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Bladder (Renal and urinary disorders) | 2 (2)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Head/headache (Nervous system disorders) | 1 (1)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other: Headache (Nervous system disorders) | 1 (3)
Pain - Other: Oral Cavity (Gastrointestinal disorders) | 1 (1)
Pain - Pain NOS (General disorders) | 1 (1)
Pain - Vagina (Reproductive system and breast disorders) | 1 (1)
Personality/behavioral (Psychiatric disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (8)
Proteinuria (Renal and urinary disorders) | 1 (2)
Pulmonary/Upper Respiratory - Other: Rhinorrhea (Infections and infestations) | 1 (2)
Pulmonary/Upper Respiratory - Other: Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (6)
Rigors/chills (General disorders) | 2 (2)
Sexual/Reproductive Function - Other: Menstrual cramps (Reproductive system and breast disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 (15)
Supraventricular and nodal arrhythmia - Sinus arrhythmia (Cardiac disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes